CLINICAL TRIAL: NCT04997967
Title: Ketofol Versus Propofol in Urgent ERCP for Acute Cholangitis: A Randomized Controlled Trial
Brief Title: Ketofol Versus Propofol in Urgent ERCP for Acute Cholangitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidi Karam, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Ketofol in Urgent ERCP
Record Dates: First submitted 2021-07-11; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Conscious Sedation Failure During Procedure
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketofol group (Experimental): Patients undergoing urgent therapeutic ERCP for severe cholangitis, with American Society of Anaesthesiologist (ASA) Grade II - III. Will receive Ketofol (ketamine: propofol concentration 1:4) prepared in 50 ml syringe containing dextrose 5% (each ml contained 8 mg propofol and 2 mg ketamine), administered as following; 5 ml of ketofol as loading then infusion titrated till targeted RSS score.
  Interventions: Drug: Ketamine/Propofol
- Propofol group (Active Comparator): Patients undergoing urgent therapeutic ERCP for severe cholangitis, with American Society of Anaesthesiologist (ASA) Grade II - III. Sedation was initially started by bolus dose of 0.5 mg/kg propofol IV over 3 minutes then, infusion was started at the rate of 50 µg /kg/min till RSS score of 5.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine/Propofol — The level of sedation was assessed at 1-3 min intervals, and the infusion rate was adjusted accordingly to achieve a Ramsay Sedation Scale (RSS) score of 5. Any movement of the patient was treated by increasing infusion rate and the infusion was discontinued at the end of the procedure. The total propofol consumed was calculated and the recovery time was recorded and calculated as the time from discontinuation of infusion of the study drug till achievement of RSS score of 3. Then patients were discharged to post-anesthesia care unit (PACU) after attaining an Aldrete Recovery Scale Score of 9- 10 [19]. Time taken to achieve this score was also recorded.
  Arms: Ketofol group
Drug: Propofol — Sedation was initially started by bolus dose of 0.5 mg/kg propofol IV over 3 minutes then, infusion was started at the rate of 50 µg /kg/min till RSS score of 5.
  Arms: Propofol group

SUMMARY:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is a lengthy and uncomfortable procedure that requires adequate sedation. Propofol is the commonly used sedative during ERCP. However, dose dependent cardiac and respiratory depression may occur. Hypotension usually occurs in severe cholangitis which necessitate the use of alternative sedative. The aim is to study the efficacy and safety of ketofol as a sedative during urgent ERCP for severe cholangitis.

DETAILED DESCRIPTION:
This randomized controlled trial was carried out on 96 patients undergoing urgent ERCP for severe cholangitis. Patients were allocated into two groups; group 1: received ketofol and group 2: received propofol. Demographic data, ERCP duration, recovery time, heart rate (HR), mean arterial pressure (MAP), peripheral oxygen saturation, Ramsey Sedation Scale (RSS), pain Numerical Rating Scale (NRS), propofol requirement, adverse events, endoscopists and patients satisfaction were recorded

ELIGIBILITY:
Inclusion Criteria:

* Severe acute cholangitis of either sex
* Aged between 21-70 years
* Undergoing urgent therapeutic ERCP for severe cholangitis with American Society of Anaesthesiologist (ASA) Grade II - III.

Exclusion Criteria:

* Patients who had ASA physical status Grade VI,
* Baseline SpO2 <90%,
* Patients who had difficulty in communication,
* Patients allergic to the studied medications,
* Morbidly obese patients,
* Patients with chronic obstructive pulmonary disease,
* Complicated airway,
* Pregnant patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ketofol in sedation | 24 hours
  The time to reach Ramsay Sedation Scale score of 5 to ensure adequate sedation. This scale is between 1-6.
  The score 5 and 6 indicates adequate sedation while score <5 indicates inadequate sedation.

SECONDARY OUTCOMES:
Impact of ketofol on hemodynamics | 24 hours
  Heart rate (beats/min)
Impact of ketofol on oxygen saturation | 24 hours
  Pulse oximeter (SO2)
Impact of ketofol on hemodynamics | 24 hours
  Blood pressure(mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Haidi Ramadan, PhD, Principal Investigator — faculty of medicine
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Direct contact with the PI